CLINICAL TRIAL: NCT06415734
Title: Repeated Transcranial Magnetic Stimulation (rTMS) Promotes Neural Function Recovery in Patients With Ischemic Stroke by Affecting Local Cerebral Blood Flow and Brain Network
Brief Title: Effect of Repetitive Transcranial Magnetic Stimulation on Neurological Recovery in Patients With Ischaemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202405n
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Stroke Ischemic
Keywords: rTMS; stroke Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (Experimental): Subjects were treated with transcranial magnetic stimulation with the addition of a figure-of-eight coil on top of conventional western medicine treatment, and the treatment modalities were all LF-rTMS 20 min, 1200 pulses, 120% RMT in M1 contralateral to the brain lesion, with a treatment cycle of 5 days. And subjects will be assessed on the relevant scales on Day 1 and Day 5 of treatment and will be tested using a near infrared functional brain imaging device before, during and after treatment on that day.
  Interventions: Device: rTMS
- control (No Intervention): Patients received only conventional Western medications. And subjects will be assessed on the relevant scales on Day 1 and Day 5 of treatment and will be tested using a near infrared functional brain imaging device before, during and after treatment on that day.

INTERVENTIONS:
Device: rTMS — LF-rTMS of M1 contralateral to the brain lesion for 20 min, 1200 pulses, 120% RMT, treatment cycle of 5 days
  Arms: rTMS

SUMMARY:
The goal of this clinical trial is to learn if transcranial magnetic stimulation(rTMS) can improve neurological rehabilitation in patients with acute ischemic stroke. The main questions it aims to answer are:

Can rTMS Promote Recovery of Limb Impairment in Patients with Acute Ischemia? Can rTMS Cause Changes in the Functional Connections of Brain Networks in Patients?

Researchers will compare rTMS therapy to non-stimulation therapy to see if rTMS is effective in promoting neurological recovery from ischemic stroke.

Participants will:

Receive rTMS or sham stimulation with LF-rTMS on the contralateral M1 of the brain lesion for 20 minutes, 1200 pulses, 120% RMT, and a treatment period of 5 days； Be evaluated on a scale before and after treatment

ELIGIBILITY:
Inclusion Criteria:

1. The age range is 18~75 years old
2. Meet the diagnostic criteria of China Acute Ischaemic Stroke Diagnosis and Treatment Guidelines 2018 and confirmed by head CT or MRI scanning
3. Acute stage of the disease <14 days and stable condition
4. Stroke patients with only unilateral limb involvement (without bilateral cerebrovascular lesions)
5. Patients with upper limb muscle strength ≥ grade 3, able to perform fNIRS tasks with the patient.
6. Subjects were right-handed
7. Participants give their informed consent and sign an informed consent form

Exclusion Criteria:

1. Those who have metal implants or any electronic devices in their body
2. Those with previous epilepsy or mental abnormality.
3. Combined with serious heart, liver, lung and other important organ failure
4. Those who have brain haemorrhage or bleeding tendency.
5. Deteriorating condition, new cerebral infarction or secondary cerebral haemorrhage.
6. Patients with history of craniocerebral trauma and craniocerebral surgery.
7. Those with severe cognitive and communication disorders who are unable to cooperate -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in patient motor function | Before patient treatment and 5 days after patient treatment
  Fugl-Meyer assessment scale，FMA Score: Minimum: 0 points, Maximum: 100 points The higher the score, the better the limb function.

SECONDARY OUTCOMES:
Altered functional connectivity of brain networks in patients | Patient before and after treatment on the first and fifth day of treatment and during rTMS treatment
  data from near-infrared functional brain imaging acquisitions

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF